CLINICAL TRIAL: NCT00989352
Title: Treatment of Patients Over 65 Years With Primary CNS Lymphoma: High-dose Methotrexate Combined With Chemo-immunotherapy Followed by Maintenance Therapy
Brief Title: Methotrexate-based Chemo-immunotherapy Followed by Maintenance Therapy for Patients > 65 Years With Central Nervous System (CNS)-Lymphoma
Acronym: PRIMAIN
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Freiburg (Other)
Collaborators: Universitätsklinikum Köln (Other); Ludwig-Maximilians - University of Munich (Other); University Hospital Heidelberg (Other); University Hospital Ulm (Other)
Responsible Party: PD Dr. Gerald Illerhaus,, University Medical Center Freiburg, Dept. of Internal Medicine I - Hematology and Oncology
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00591; Eudract: 2008-007645-31
Record Dates: First submitted 2009-10-02; First posted 2009-10-05 (Estimated); Last update posted 2009-10-05 (Estimated); Status verified 2009-10

CONDITIONS: Primary Non Hodgkin Lymphoma of the Central Nervous System
Keywords: PCNSL; Lymphoma; Methotrexate; Lomustine; Procarbazine; Rituximab; Elderly; Chemotherapy
MeSH Terms: conditions — Lymphoma | interventions — Methotrexate; Lomustine; Procarbazine; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Methotrexate — 3g/m² i.v. max. 9 times
Drug: Lomustine — 110 mg/m² p.o., max. 3 times
Drug: Procarbazine — 60 mg/m² p.o. for 10 days, max. 3 times 100 mg p.o. for 5 days, max. 6 times
Drug: Rituximab — 375 mg/m² i.v., max. 10 times

SUMMARY:
The purpose of this study is to determine whether combined chemotherapy [rituximab plus high dosage methotrexate, lomustine, and procarbazine] followed by maintenance therapy with procarbazine is effective in the treatment of cerebral Non Hodgkin lymphoma [PCNSL] in patients > 65 years.

ELIGIBILITY:
Inclusion Criteria:

* first diagnosis of PCNSL, histologically confirmed
* age > 65 years
* written signed and dated informed consent of the legal representative and - if possible - of the patient

Exclusion Criteria:

* manifestations of further lymphoma outside the CNS
* sero-positive for HIV
* severe pulmonary, cardiac, hepatic, renal impairment
* uncontrolled infection
* neutrophil count < 1.500/µl, platelet count < 100.000/µl
* pulmonary disease with IVC < 55%, DLCO < 40%
* cardiac ejection fraction < 50%, uncontrolled malign arrhythmia
* creatinine > 1,5 mg% or creatinine-clearance < 50ml/min
* bilirubin > 2mg/dl
* ascites or pleural effusion (> 500ml)
* known hypersensitivity against methotrexate, lomustine, procarbazine, rituximab, leukovorin, or dexamethasone
* participation in another clinical trial within the last 30 days prior to the begin or parallel to this study
* known or current drug or alcohol abuse

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-06 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate | 30 days after end of immuno-chemotherapy

SECONDARY OUTCOMES:
Duration of response | within 5 years
Overall survival time | within 5 years
Neuropsychological state (according to Mini-Mental State and IPCG testing) | within 5 years
(Serious) adverse events ([S]AEs) | within 30 days after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Illerhaus, PD Dr., Principal Investigator — University Medical Center Freiburg, Dept. of Internal Medicine I - Hematology and Oncology
Locations (1):
- University Medical Center Freiburg, Dept. of Internal Medicine I - Hematology and Oncology, Freiburg im Breisgau, Germany

REFERENCES:
- [Background] Illerhaus G, Marks R, Muller F, Ihorst G, Feuerhake F, Deckert M, Ostertag C, Finke J. High-dose methotrexate combined with procarbazine and CCNU for primary CNS lymphoma in the elderly: results of a prospective pilot and phase II study. Ann Oncol. 2009 Feb;20(2):319-25. doi: 10.1093/annonc/mdn628. Epub 2008 Oct 26. PMID 18953065
- [Derived] Fritsch K, Kasenda B, Schorb E, Hau P, Bloehdorn J, Mohle R, Low S, Binder M, Atta J, Keller U, Wolf HH, Krause SW, Hess G, Naumann R, Sasse S, Hirt C, Lamprecht M, Martens U, Morgner A, Panse J, Frickhofen N, Roth A, Hader C, Deckert M, Fricker H, Ihorst G, Finke J, Illerhaus G. High-dose methotrexate-based immuno-chemotherapy for elderly primary CNS lymphoma patients (PRIMAIN study). Leukemia. 2017 Apr;31(4):846-852. doi: 10.1038/leu.2016.334. Epub 2016 Nov 15. PMID 27843136
- See also: Related Info — http://www.zns-lymphome.de